CLINICAL TRIAL: NCT04090788
Title: The Effect of Momordica Charantia Supplementation on Blood Glucose Levels
Acronym: Bitter-sweet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University and Research (Other)
Responsible Party: Principal Investigator, Diederik Esser, Project leader clinical trials, Wageningen University and Research
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NL70259.081.19
Record Dates: First submitted 2019-09-10; First posted 2019-09-16 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2019-09

CONDITIONS: Glucose Intolerance
Keywords: bitter gourd; pre-diabetics; glucose response
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dried bitter-gourd supplements (Experimental): 2.4 gram per day for 4 weeks
  Interventions: Dietary Supplement: dried bitter-gourd supplements
- dried cucumber supplements (Active Comparator): 2.4 gram per day for 4 weeks
  Interventions: Dietary Supplement: dried cucumber supplements

INTERVENTIONS:
Dietary Supplement: dried bitter-gourd supplements — intervention with 2.4g/d dried bitter-gourd supplements
  Other Names: Momordica charantia
  Arms: dried bitter-gourd supplements
Dietary Supplement: dried cucumber supplements — reference intervention with 2.4g/d dried cucumber supplements
  Arms: dried cucumber supplements

SUMMARY:
The study is a randomized, cross-over, double blind, controlled trial in which study participants will receive two 4-week interventions with a washout period of 4 weeks between interventions. Study subjects will visit the research facility before and after each intervention period for a test day. In the third intervention week participants are provided with a 3-day controlled diet and glucose responses will be monitored via a continuous glucose monitoring device.

DETAILED DESCRIPTION:
Bitter gourd (BG) (Momordica charantia), is a highly nutritive vegetable from the cucumber family. The objective is to assess the impact of 4-week BG supplementation on blood glucose levels and glucose tolerance in subjects with an impaired fasting glucose or with an impaired glucose tolerance and to evaluate how BG supplements modulate glucose response curves during meal intake. The study is a randomized, cross-over, double blind, controlled trial in which study participants will receive two 4-week interventions with a washout period of 4 weeks between interventions. Study subjects will visit the research facility before and after each intervention period for a test day. In the third intervention week participants are provided with a 3-day controlled diet and glucose responses will be monitored via a continuous glucose monitoring device. The intervention will be a 4-week intervention with 2.4g/d dried bitter-gourd supplements and a reference intervention with 2.4g/d dried cucumber supplements. The main study parameter is fasting levels of plasma glucose and 2hour plasma glucose after a 75-gram OGTT.

ELIGIBILITY:
Inclusion Criteria:

* age 50-75yrs
* BMI >25 kg/m2
* Having veins suitable for blood sampling via a catheter
* Having one or more of the following criteria:

  * HbA1c > 5.7%
  * fasting glucose >5.6mmol/L
  * two-hour glucose levels >7.8 mmol/L on the 75-g oral glucose tolerance test .

Exclusion Criteria:

* History of gastro-intestinal surgery or having (serious) gastro-intestinal complaints
* History of liver dysfunction (cirrhosis, hepatitis) or liver surgery
* Kidney dysfunction (self-reported)
* Use of medication/supplements that may influence the study results, such as medicines known to interfere with glucose homeostasis.
* Anaemia (Hb values <7.5 for women and <8.5 for men)
* Reported slimming, medically prescribed or other extreme diets
* Reported weight loss or weight gain of > 5 kg in the month prior to pre-study screening
* Not willing to give up blood donation during the study
* Current smokers
* Alcohol intake ≥4 glasses of alcoholic beverages per day
* Abuse of illicit drugs
* Food allergies for products that we use in the study
* Participation in another clinical trial at the same time
* Being an employee of the Food, Health & Consumer Research group of Wageningen Food & Biobased Research or dept. human nutrition and health of Wageningen University.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2019-12-24 (Actual); Study Completion 2019-12-25 (Actual)

PRIMARY OUTCOMES:
change in fasting plasma glucose concentrations | before (Week 0) and after 4 weeks of supplement intervention
  marker for glucose metabolism
change in 2hour plasma glucose concentrations after a 75-gram OGTT | before (Week 0) and after 4 weeks of supplement intervention
  marker for glucose metabolism

SECONDARY OUTCOMES:
change in HbA1c | before (Week 0) and after 4 weeks of supplement intervention
  marker for glucose metabolism
change in fructosamine | before (Week 0) and after 4 weeks of supplement intervention
  marker for glucose metabolism
change in fasting insulin | before (Week 0) and after 4 weeks of supplement intervention
  marker for glucose metabolism
change in 2hour plasma insulin concentrations after a 75-gram OGTT | before (Week 0) and after 4 weeks of supplement intervention
  marker for glucose metabolism
Change in postprandial glucose concentrations after food intake | Three full days, in the third week of the supplement intervention
  measured by a continues glucose monitoring device

OTHER OUTCOMES:
change in triglycerides (TAG) concentration | before (Week 0) and after 4 weeks of supplement intervention
  marker of lipid metabolism
change in cholesterol | before (Week 0) and after 4 weeks of supplement intervention
  marker of lipid metabolism
change in ALAT | before (Week 0) and after 4 weeks of supplement intervention
  Liver enzyme
change in ASAT | before (Week 0) and after 4 weeks of supplement intervention
  Liver enzyme
change in eGFR (CKD-EPI) | before (Week 0) and after 4 weeks of supplement intervention
  Liver enzyme

CONTACTS AND LOCATIONS:
Locations (1):
- Stichting Wageningen Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No